CLINICAL TRIAL: NCT05440240
Title: Percutaneous Needle Fasciotomy (PNF) +/- Corticosteroid Injection for Dupuytren's Contracture (DC) Affecting Metacarpophalangeal Joints (MCP) . A Randomized Controlled Trial
Brief Title: Percutaneous Needle Fasciotomy +/- Corticosteroid Injection for Dupuytren's Contracture
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Laura Houstrup Matthiesen, Medical Student, PhD Student, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-985; 2022-501021-20-00 (Other: EU CT)
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Dupuytren Contracture; Dupuytren's Disease; Contracture; Joint Diseases; Musculoskeletal Diseases; Fibroma; Neoplasm, Fibrous Tissue; Neoplasms, Connective Tissue; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms; Connective Tissue Diseases
Keywords: Percutaneous needle fasciotomy; Corticosteroid; Randomized controlled trial
MeSH Terms: conditions — Dupuytren Contracture; Contracture; Joint Diseases; Musculoskeletal Diseases; Fibroma; Neoplasms, Fibrous Tissue; Neoplasms, Connective Tissue; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms; Connective Tissue Diseases | interventions — Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid injection (Active Comparator): Percutaneous needle fasciotomy with corticosteroid injection
  Interventions: Procedure: Percutaneous needle fasciotomy; Drug: Corticosteroid injection
- Saline injection (Placebo Comparator): Percutaneous needle fasciotomy with saline injection
  Interventions: Procedure: Percutaneous needle fasciotomy; Other: Saline injection

INTERVENTIONS:
Procedure: Percutaneous needle fasciotomy — Percutaneous needle fasciotomy ad modum Lermusiaux and Debeyre
Drug: Corticosteroid injection — Depo-Medrol
  Arms: Corticosteroid injection
Other: Saline injection — Isotonic saline
  Arms: Saline injection

SUMMARY:
Comparing percutaneous needle fasciotomy +/- corticosteroid injection for Dupuytren's contracture affecting metacarpophalangeal joints. A clinician-initiated, multicenter, randomized controlled trial.

ELIGIBILITY:
Sufficient correction of metacarpophalangeal (MCP) joint during the PNF treatment, defined as <20° passive extension deficit (PED), is a prerequisite for inclusion.

Inclusion Criteria:

* Dupuytren contracture (DC) of ≥ 20° PED in MCP joint measured with a goniometer
* DC of either II-V finger
* Well-defined/palpable cord

Exclusion Criteria:

* Legally incapacitated
* Previous study inclusion with another finger ray
* Isolated proximal interphalangeal (PIP) or distal interphalangeal (DIP) joint contracture, defined as MCP joint contracture < 20° PED regardless of the deficit in the PIP or DIP joint
* Previous hand surgery of the affected finger for any reason
* Known allergy to the study medication
* Anticoagulant therapy (Acetylsalicylic acid is NOT an exclusion criterion)
* Pregnant or lactation
* Insulin dependent diabetes mellitus
* Ongoing systemic infection or local infection at the site of the procedure
* Rheumatoid arthritis
* Amyloidosis or mucopolysaccharidosis
* Unable to communicate, cooperate or participate in follow-up

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years
  Recurrence is defined as 20 degrees or more passive extension deficit in metacarpophalangeal joint from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Lange, MD, PhD, Study Director — Regionshospitalet Horsens
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matthiesen LH, Skov ST, Lange J. Adjuvant steroid to percutaneous needle fasciotomy for Dupuytren's contracture. An RCT study protocol. Dan Med J. 2024 Nov 12;71(12):A05240324. doi: 10.61409/A05240324. PMID 39749555